CLINICAL TRIAL: NCT01986205
Title: A Double-blind Randomized Trial of Hyperbaric Oxygen Versus Sham for Persistent Symptoms After Brain Injury
Brief Title: Hyperbaric Oxygen for Traumatic and Non-traumatic Brain Injury
Acronym: HYBOBI2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lindell Weaver (Other)
Responsible Party: Sponsor-Investigator, Lindell Weaver, Medical Director, Hyperbaric Medicine, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1024845
Record Dates: First submitted 2013-10-31; First posted 2013-11-18 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Brain Injury, Chronic
Keywords: Concussion; Traumatic brain injury; Hyperbaric oxygenation; Post-concussion symptoms; Headache; Carbon monoxide
MeSH Terms: conditions — Brain Injury, Chronic; Brain Concussion; Brain Injuries, Traumatic; Post-Concussion Syndrome; Headache | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hyperbaric Oxygen (Experimental): 100% oxygen at 1.5 atmospheres absolute for 60 minutes, 40 sessions
  Interventions: Combination Product: Hyperbaric Oxygen
- Minimal pressure air (Placebo Comparator): Regular air at minimal pressurization for 60 minutes, 40 sessions
  Interventions: Combination Product: Minimal pressure air

INTERVENTIONS:
Combination Product: Hyperbaric Oxygen — Hyperbaric oxygen (USP oxygen >99%) delivered in a hyperbaric chamber pressurized to 1.5 atmospheres absolute.
  Other Names: HBO2; HBOT; HBO; Hyperbaric oxygen therapy
  Arms: Hyperbaric Oxygen
Combination Product: Minimal pressure air — Room air delivered in a hyperbaric chamber with minimal pressurization.
  Other Names: Room air
  Arms: Minimal pressure air

SUMMARY:
The purpose of this study is to examine whether 40 hyperbaric oxygen sessions has effect on long-term symptoms after brain injury. This study will enroll 90 individuals with persistent problems 6 months to 10 years after a brain injury. These individuals will be randomized to receive either oxygen or air in a pressurized hyperbaric chamber. Participants will receive 40 daily hyperbaric chamber sessions.

Participants will have a series of tests and questionnaires before they begin their chamber sessions, after they complete 40 sessions, and 6 months after they joined the study. These tests include computer-based and pencil-and-paper questionnaires and thinking tests, brain imaging, a neurological examination, and an eye exam. Participants will also be asked to provide blood for future research.

After the 6-month tests are complete, all participants will receive 40 hyperbaric oxygen sessions, then undergo the same tests at 9 months and 12 months.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind study with a subsequent open-label intervention period to explore whether a course of hyperbaric oxygen can ameliorate persistent symptoms after brain injury. In this study, adult men and women with persistent symptoms 6 months to 10 years after injury will be randomized to receive 40 hyperbaric oxygen sessions (100% oxygen at 1.5 atmospheres absolute, 60 minutes door-to-door) or sham chamber sessions (room air chamber excursion at near-ambient pressure, 60 minutes door-to-door). Chamber sessions will be provided Monday through Friday, excluding holidays, and participants will have up to 12 weeks to complete their 40 sessions.

Participants will be evaluated before the chamber sessions, at 13 weeks, and at 6 months. Assessments include self-administered questionnaires, neuropsychological function, a brief neurological examination, electroencephalography, visual function tests, and a neuro-optometry evaluation. These outcome tools will measure symptoms and deficit at the time of enrollment and subsequent evaluations, and provide insight into whether hyperbaric oxygen can play a role in recovery from brain injury.

Once the participants have completed their 6 month evaluations, they will enter an open intervention group, receiving 40 hyperbaric sessions at 1.5 atmospheres absolute for 60 minutes. Participants will have up to 12 weeks to complete these sessions. Participants will be evaluated after the second set of chamber sessions (at 9 months and again at 12 months). Individuals will then be assessed annually until study closure (12-month follow-up of the last enrolled participant).

Participants will be asked to provide blood for long-term storage of serum, plasma, and DNA for future investigations, including apolipoprotein E genotype.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18-70 years, both men and women
* Able to speak and read English as primary language
* Able and willing to provide written informed consent for study participation.
* Able and willing to complete outcome assessments and provide blood and urine samples as required by the study protocol.
* Able to tolerate the chamber environment and hood placement and to equalize middle ear pressure.
* Past history of at least one brain injury with persistent symptoms that meets all of the following criteria:

  * Brain injury of non-stroke etiology that occurred at least 6 months but no more than 10 years prior to enrollment.
  * At least 3 of the following persistent symptoms from the injury: headaches, dizziness or balance problems, blurred vision, tiredness/fatigue or sleep problems, seizures, remembering things or solving problems, managing stress or emotional upsets, controlling temper/irritability, depression, anxiety, post-traumatic stress, or ringing in the ears.
* Normal thyroid stimulating hormone and hematocrit value greater than 35% within the previous 6 months.

Exclusion Criteria:

* Contraindications to hyperbaric oxygen

  * Insulin-dependent diabetes mellitus, or diabetes mellitus that is not reasonably controlled.
  * Uncontrolled seizure disorder (participants must be on therapy and seizure-free for at least 6 months).
  * Claustrophobia precluding chamber or hood tolerance.
  * Implanted devices not cleared for hyperbaric pressurization.
  * Pregnancy or plans to become pregnant during the study participation period. Women of childbearing potential will be asked to use an acceptable form of birth control during study participation.
  * Lung disease, such as emphysema, chronic bronchitis, asthma that is not well-controlled, or bullous lung disease that raises the risk for pulmonary barotrauma due to air trapping.
  * Active malignancy, previous malignancy (except basal cell carcinoma) in the last 5 years, or any prior treatment with bleomycin (Blenoxane). Prior treatment with doxorubicin (Adriamycin) is acceptable as long follow-up echocardiography is normal.
  * Chronic disease such as heart or renal failure would raise the participant's risk of adverse events during hyperbaric oxygen.
* Confounds to the outcome assessments

  * Inability to speak English as their primary language (English fluency required because many of the outcomes are only in available in English)
  * Instability with walking requiring more than a cane for assistance
  * Alcohol abuse, by self-report, within the last year.
  * Lifetime history of illicit drug use, by self-report, except remote (greater than one year), non-habitual use of marijuana.
  * Failed urine drug screen during study participation.
  * Continued participation during the intervention period in sports activities where head injury is likely, such as contact football, boxing, mixed martial arts, etc.
  * Blind or deaf.
  * Major psychiatric disorder or degenerative mental disease (such as multiple sclerosis).
  * Prior therapeutic radiation to the central nervous system.
  * Personal history of any condition that pre-dates their brain injury that resulted in diminished capacity (such as chromosomal disorders) or that, in the opinion of the investigators, affects cognition to such a degree that the outcome assessments are invalidated (such as learning disability or attention deficit hyperactivity disorder requiring pharmaceutical therapy as an adult).
  * Any brain injury from stroke (ischemic or hemorrhagic)
  * Known untreated chronic or acute medical conditions, such as hypothyroidism, Cushing's disease, untreated hypertension, etc., that would confound the outcome assessments or inhibit compliance with the study protocol. If treated, these disorders would not be excluded.
  * Concomitant enrollment in any other drug/device clinical trial.
  * Prior hyperbaric oxygen for any reason within the last year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Neurobehavioral Symptom Inventory | 13 weeks
  Participant-reported symptom rating of post-concussive symptoms

SECONDARY OUTCOMES:
Neurobehavioral Symptom Inventory | 6 months
  Participant-reported symptom rating of post-concussive symptoms
Incidence of myopia | 13 weeks
  Myopic visual changes after chamber sessions

CONTACTS AND LOCATIONS:
Overall Officials: Lindell K. Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - Intermountain LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Churchill S, Weaver LK, Deru K, Russo AA, Handrahan D, Orrison WW Jr, Foley JF, Elwell HA. A prospective trial of hyperbaric oxygen for chronic sequelae after brain injury (HYBOBI). Undersea Hyperb Med. 2013 Mar-Apr;40(2):165-93. PMID 23682548